CLINICAL TRIAL: NCT07090915
Title: Evaluating the Impact of Nature Soundscapes on Post-Operative Stress and Anxiety in Orthopedic Surgery Patients
Brief Title: The Influence of Natural Sounds on the Well-being of Patients After Orthopaedic Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Michael Tobias Hirschmann (Other)
Responsible Party: Sponsor-Investigator, Michael Tobias Hirschmann, Prof. Dr. med., Kantonsspital Baselland Bruderholz
Organization: Kantonsspital Baselland Bruderholz (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2025-01087
Record Dates: First submitted 2025-06-27; First posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Postoperative Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): standard hospital stay
- Intervention group (Experimental)
  Interventions: Other: nature sound

INTERVENTIONS:
Other: nature sound — Modern audio technology is used to create a 3D natural atmosphere.
  Arms: Intervention group

SUMMARY:
For many people, a stay in hospital can be associated with stress and anxiety, especially after surgery. In order to potentially make the stay more pleasant for patients in future, the investigators are conducting a study to investigate the use of natural sounds to promote relaxation. Participation in this study usually lasts until 3 days after the operation in hospital. If the participants decide to take part, the participants will be randomly assigned to one of two groups: The intervention group or the control group. In the intervention group, the participants will listen to different natural sounds twice a day. In the control group, the participants will not receive any nature sounds. During the stay, the participants will be given two questionnaires to fill in about how you feel. Participants assigned to the intervention group will additionallyreceive a short telephone interview 14 days after the operation.

ELIGIBILITY:
Inclusion Criteria:

1. duly completed declaration of consent
2. the age of the patient is at least 18 years
3. only patients undergoing orthopaedic surgery

Exclusion Criteria:

1. deafness
2. severe cognitive impairment
3. chronic pain patient
4. pain catheter insertion during the trial period
5. psychiatric disorders (e.g. anxiety disorders, depression, post-traumatic stress disorder, ...)
6. severe postoperative complications
7. no consent to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Depressions-Angst-Stress-Skalen (DASS-21) | From the first day after surgery until the third day after surgery.
  0 to 63 (0 is best 63 is bad)

SECONDARY OUTCOMES:
Relaxation State Questionnaire (RSQ), to measure the Relaxation | From the first day after the surgery to the third day after the surgery.
  10 to 50 (10 is not relaxed, 50 is most relaxed)
NRS, to measure the Painlevel | From the first day after the surgery to the third day after the surgery.
  0 to 10 (0 is no pain, 10 is most pain)
NRS, to measure the sleep quality | From the first day after the surgery to the third day after the surgery.
  0 to 10 (0 is no sleep, 10 ist best sleep)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Hirschmann, Prof. Dr. med., Principal Investigator — Universitäres Zentrum Bewegungsapparat, Kantonsspital Baselland Bruderholz
Locations (1):
- Universitäres Zentrum Bewegungsapparat, Kantonsspital Baselland Bruderholz, Basel, Bruderholz, Germany

IPD SHARING:
Plan to Share IPD: No